CLINICAL TRIAL: NCT06150261
Title: Tolerability and Effects of a New Omega-3 Fatty Acid-based Supplement on Clinical and Biological Markers of Healthy Ageing
Brief Title: Effects of an Omega-3 Fatty Acid-based Supplement on Healthy Ageing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Evonik Industries AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AvailOm
Record Dates: First submitted 2023-09-07; First posted 2023-11-29 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-05

CONDITIONS: Healthy Aging; Ageing Well

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind placebocontrolled, paralell-group trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AvailOm (Experimental): Availom capsules will be administered orally in a dose of 5 capsules/day per individum for a total of 6 months.
  Interventions: Dietary Supplement: AvailOm
- Placebo (Placebo Comparator): Placebo capsules matching AvailOm will be administered orally in a dose of 5 capsules/day per individum for a total of 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AvailOm — 5 capsules taken once daily with main meal
  Arms: AvailOm
Dietary Supplement: Placebo — 5 capsules taken once daily with main meal
  Arms: Placebo

SUMMARY:
The goal of this randomised, double-blind placebo controlled trial is to explore tolerability and the effects of a new omega-3 fatty acid-based supplement on biological and clinical aspects relevant for healthy ageing.

Participants will be asked to take a supplement or a placebo for 6 months, and to attend the clinic a total of 3 times and to perform or submit the following:

* Physical examination
* Muscle function tests
* Cognitive testing
* Questionnaire completion
* Biological samples, including blood, saliva and faeces.

Researchers will compare the results from the group taking the supplement to the results of the group taking a placebo to see if the supplement has an effect on biological and clinical aspects associated with healthy ageing.

DETAILED DESCRIPTION:
Healthy ageing is the process of developing and maintaining the functional ability that is associated with wellbeing across the life course and comprises mental and physical capacities such as the ability to walk, think, see, hear and remember. These factors are influenced by several factors including diseases, age-related decline in organ function and lifestyle such as diet and physical exercise.

Among dietary factors, omega-3 fatty acids, including eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), are increasingly recognized as potentially promoting healthy ageing, including benefits to cardiovascular system, as well as muscle function, and brain function. It is also important for brain and eye development. Regular supplementation with EPA and DHA therefore potentially offers a range of health benefits throughout life.

Since humans cannot synthesize omega-3 fatty acids, these are considered essential nutrients and must be incorporated into the diet, with the main source for EPA and DHA incorporation being fish oils and supplementation. Western diets are often deficient in these compounds, therefore, regular supplementation with EPA and DHA potentially delays functional decline in ageing and reduces the incidence / severity of age-related diseases.

Objective/Aims:

Explore tolerability and the effects of the IP on biological and clinical aspects relevant for healthy aging.

Design:

Randomized, double-blind placebo-controlled parallel-group trial for six months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55 or more
* BMI between 25-30,
* Waist-to-hip ratio of at least 0.90 (males) or 0.85 (females)
* Omega-3 index <6

Exclusion Criteria:

* Dementia
* Current clinically significant depression, i.e. major depression or GDS 15 score >7
* Ischemic or haemorrhagic Stroke
* Acute myocardial infarction
* Any form of clinically significant atherosclerotic cardiovascular disease
* Unstable angina pectoris
* Hearth failure in need of treatment
* Diabetes mellitus type 1 or 2
* Clinically relevant kidney diseases that require dialysis, including clinically significant chronic kidney disease
* Liver cirrhosis or active hepatitis B or C
* Cancer of any kind; however, benign tumours are no exclusion criterium
* Clinically relevant inflammatory or autoimmune disorders with history of hospitalisation
* Any form of systemic lupus erythematosus (SLE), rheumatoid arthritis, Colitis ulcerosa, Crohn's disease, Morbus Parkinson, Multiple Sclerosis
* hsCRP > 3.0 mg/L to exclude high risk individuals according to international criteria
* LDL-C > 160mg/dL to exclude individuals with high risk for arterioscleratic coronary disease26
* HBa1C < 6.5% to exclude diabetes
* Fasting Triglycerides >200 mg/dL
* Omega 3 index > 6 % (as they may not show any benefit from supplementation)
* Use of fish oil / omega 3 supplements over the last 6 months
* Fish allergy
* Antibiotic use in the last 24 weeks

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effects of Availom on DNA methylation | 6 months
  Effects of Availom on DNA methylation will be measured by a novel saliva-based method and correlated with the individual's genotype. EPIC (850k) chip platform for DNA methylation patterns will be used to measure these changes.

SECONDARY OUTCOMES:
Effects of Availom on inflammation | 6 months
  Blood will be analysed for markers of inflammation (CRP and cytokines; eg TNFa, IL6), using commercially available immunoassays all measurements will be in pg/ml.
Effects of Availom on plasma lipids | 6 months
  Changes in plasma lipids will be measured; Omega-3 fatty acids and their metabolites, especially eicosanoids, resolvins D1, EPA/DHA levels, LDL-cholesterol. Commercially available immunoassays will be used. The unit of measurement for all measures will be pg/ml.
Effects of Availom on in vitro neurogenesis markers | 6 months
  Serum obtained from participants at baseline and end point visit will be used to treat hippocampal progenitor cells in an established in vitro model of hippocampal neurogenesis, developed by the Thuret lab at KCL. This will be an entirely in vitro experiment using only the serum samples from this trial's participants.
  Following cell culture and immunocytochemistry, this assay provides information on the neurogenic potential of each individual. Neurogenic potential is measured as percentage cells positive for SOX2/ NESTIN/ KI67/ CC3 /DCX and MAP2.
  The values obtained from cells treated with endpoint samples will be compared to values obtained from cells treated with baseline samples for each individual to control for inter-individual differences allowing us to use this set up to establish if 6 months of availom can alter an individuals neurogenic potential.
Effects of Availom on brain-derived neurotrophic factor | 6 months
  Levels of BDNF has been shown to be a reliable index as biomarker for assessing the effectiveness of Omega-3 supplements in improving brain function.
Effect of Availom on microbiome changes | 6 months
  DNA will be extracted from stool samples provided by study subjects and the microbial composition determined following next-generation sequencing to assess the effect of Availom on microbial composition.
Investigate potential moderators of the effect of Availom on microbial composition | 6 months
  Microbiome data obtained in outcome 7 will be analysed and correlated to (meta)data collected to identify key species linked to gut health.
Effects of Availom on cognition as measured by use of MoCA | 6 months
  As measured by Montreal Cognitive Assessment (MoCA). MOCA scores range between 0 and 30 points, with a higher score indicating higer cognitive function.
Effects of Availom on cognition as measured by use of CERAD | 6 months
  As measured by the word list memory test from the Consortium to establish a registry for Alzheimer's disease (CERAD) neuropsychological battery. The same list is presented in a different order three times and the participant is asked to recall as many words as possible. The maximum number of correct responses is 10 for each trial with a maximum score of 30.
Effects of Availom on muscle function as asessed by TUG | 6 months
  As measured by the Timed Up and Go test (TUG)
Effects of Availom on muscle function as assessed by grip strength | 6 months
  As measured by testing grip strength with a dynamometer
Effects of genotype on association between Availom and genotype | 6 months
  Genotype of saliva samples will be analysed using Ilumina Infinium Global Screening Array the effect of different genotypes will be assessed as a potential moderators of the association between availom and DNA methylation

CONTACTS AND LOCATIONS:
Overall Officials: Dag Aarsland, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger Universitetssjukehus, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No